CLINICAL TRIAL: NCT03468361
Title: Diuretic Effect Evaluation of Petroselinum Crispum (Parsley) in Hypertensive Patients (DEEP): Phase-I Clinical Trial
Brief Title: Diuretic Effect Evaluation of Petroselinum Crispum (Parsley) in Hypertensive Patients
Acronym: DEEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The hospitals could not enroll any patients. Therefore, the authors decided to withdraw the study.
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Atta Abbas Naqvi, Prinicipal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IAU-DEEP
Record Dates: First submitted 2018-03-11; First posted 2018-03-16 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Diurnal Enuresis; Hypertension
MeSH Terms: conditions — Diurnal Enuresis; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Patients in control group will be allowed to continue their conventional medications and with a placebo.
  Interventions: Other: Placebo
- Intervention Group (Experimental): Patients in intervention group who would be taking their usual medications along with parsley in a convenient dosage form.
  Interventions: Other: Natural Product Petroselinum crispum (Parsley)

INTERVENTIONS:
Other: Natural Product Petroselinum crispum (Parsley) — Parsley herb, in fresh form will be obtained from the local market available. The herb will be properly washed with distilled water and dried properly for 10 to 15 days under shade in the lab. Soft gelatin capsules will be filled with parsley powder (dried herb) in amount normally recommended in daily routine (1g) will be administered to patients once daily.
  Arms: Intervention Group
Other: Placebo — Soft gelatin capsules will be filled with 1 gram of lactose (inert pharmaceutical ingredient) and will be administered to patients once daily.
  Arms: Control Group

SUMMARY:
The use of alternative therapy, particularly herbal treatment is becoming prevalent among patients. Many herbs are in-use for various ailments such as diabetes, digestive problems, fever, hepatitis and hypertension etc. The common belief is, herbs are safe and easy to access as compared to conventional therapy, however, most of the studies reported different side effects which may be toxic at times. These adverse effects are mostly due to incorrect use or lack of patient education.

Parsley is a plant with antioxidant, diuretic and antimicrobial properties. Literature reported use of parsley as a diuretic by different communities in throughout the world. In vitro studies in animal have also reported the diuretic effect as well as proposed mechanisms for the use of parsley as diuretic however none of the studies have been conducted to investigate the diuretic effect of parsley in humans. This study aims to evaluate the diuretic and hence antihypertensive effect of parsley in hypertensive patients.

DETAILED DESCRIPTION:
Parsley botanically known as Petroselinum crispum, belongs to the family Umbeliferae, originated from Mediterranean region however, it is cultivated almost throughout the world now-a-days. The plant has reported folkloric uses in different parts of the world; in Iran the seeds of the plant is used for different pharmacological effects including antimicrobial, kidney stones, digestive disorders etc., in Turkey the leaves of this plant is used to treat hypertension, diabetes and as a diuretic in Morocco the leaves are used for arterial hypertension, diabetes, high blood pressure and cardiac diseases in Spain the leaves of this plant are used to treat hypertension, diabetes, prostititis and anemia whereas in Serbia the leaves of the plant are used to treat urinary tract diseases and infections. Though the aforementioned literature supports the diuretic and anti-hypertensive potential of parsley however no in-vivo studies have been reported to establish its diuretic activity in human subjects. Some studies have reported diuretic activity for seed aqueous extract in rats. Still, to evaluate the effect in human subjects, an in-vivo phase-I clinical study is needed to support the pre-clinical in-vivo and in-vitro diuretic effects of this plant. Our study aims to investigate the diuretic and anti-hypertensive activity of parsley in hypertensive individuals currently using conventional medication.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female patients with hypertension and already using conventional medications i.e. antihypertensive drugs. The consent forms will be provided to the patients and only those patients which are willing to participate will be included in the study. Patients with more than 3 co-morbidities and at high-risk conditions will not be included in the study.

Exclusion Criteria:

* Geriatric, pregnant and lactating patients will not be included in the study. More important, patients on diuretic medications as well as diabetes, will also be excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in baseline mean Blood pressure at day 7, day 14 and 21 | For observing any change in mean blood pressure, a blood pressure monitor will be used to determine any variation in blood pressure in millimeters of mercury (mm of Hg). A total of four readings will be taken at baseline day 0, day 7, day 14 and day 21.
  For observing any change in mean blood pressure, a blood pressure monitor will be used to determine any variation in blood pressure in millimeters of mercury (mm of Hg).
Change in baseline mean urinary output at day 7, day 14 and 21 | For observing any change in mean urinary output a total of four readings will be taken at baseline day 0, day 7, day 14 and day 21.
  For observing any change in mean urinary output, a urine container will be used to determine any variation in urinary output in millimeters (ml).

CONTACTS AND LOCATIONS:
Overall Officials: Dhafar M Al Shayban, PhD, Study Chair — Imam Abdulrahman Bin Faisal University; Rasha Al Sheikh, MD, Study Director — FAMCO
Locations (2):
- Saudi Arabia (2):
  - College of Clinical Pharmacy, Dammam, Eastern Province
  - FAMCO, Khobar, Eastern Province

IPD SHARING:
Plan to Share IPD: No